CLINICAL TRIAL: NCT04072783
Title: Neurodevelopmental Outcomes in Craniosynostosis Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 217610
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-12

CONDITIONS: Craniosynostoses
Keywords: Craniosynostosis; MRI; DTI; Neurodevelopment
MeSH Terms: conditions — Craniosynostoses | interventions — Diffusion Tensor Imaging; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Patients with craniosynostosis only
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients with craniosynostosis (Other): Patients with craniosynostosis will undergo pre - and post-operative imaging studies. The surgery will be performed for these patients as standard of care. They will also be tested fro neurodevelopment.
  Interventions: Diagnostic Test: MRI,DTI, functional MRI

INTERVENTIONS:
Diagnostic Test: MRI,DTI, functional MRI — 1. Patients will undergo testing with Pre- and and post-surgical MRI. The protocol will be Sagittal T1, Axial inversion recovery, T2, fluid-attenuated inversion recovery, susceptibility weighted image, diffusion weighted images, diffusion tensor imaging, resting state fMRI, sagittal 3D GRE / FFE or 3D T1 VIBE and tractography.
  2. Once patients are identified, surgery is planned.The standard of care procedures fall into two categories based on age of presentation, clinician judgement and family preference all other things being equal. Both the endoscopic-assisted craniectomy and open CVR are standard of care procedures. Patients self-select into these groups. None of the surgery nor any aspect of it is experimental.
  3. Patients are routinely examined for neurodevelopment pre- and post-operatively as part of American Cleft Palate Craniofacial Association guidelines.The Vineland Adaptive Behavior Scales are used up to and including age 4.
  Other Names: Neurodevelopmental testing, surgery

SUMMARY:
Context: Craniosynostosis is a common craniofacial abnormality which can be associated with various clinical syndromes. Though it has been established that children with craniosynostosis score lower on certain developmental tests, the effect of craniosynostosis and cranioplasty surgery on the neural circuitry and brain development is less well known or understood.

Objectives: The purpose of this study is to describe the effect of cranial vault remodeling in children with craniosynostosis on white matter tracts with tractography and Diffusion tensor imaging (DTI), functional MRI, and neurodevelopmental tests, before and after surgery as compared to age-matched controls.

Study Design: This will be a prospective study of patients diagnosed with craniosynostosis and who are going to have open or endoscopic cranial vault remodeling (CVR).

Study Measures: The study will measure MRI sequences before and after surgery and at set time intervals to quantify the effect of white matter tract maturity. Parallel to this, neurodevelopmental tests will be administered at these same intervals.

DETAILED DESCRIPTION:
Craniosynostosis, the premature ossification and fusion of one or more cranial sutures, is a common craniofacial abnormality occurring in 1 of 2,000 live births. 1 2 Craniosynostosis can lead to increased intra-cranial pressure in between 12-50% of those affected which may have delayed neuro developmental implications.

The crucial neurodevelopment occurs in the first years of life and is most rapidly progressing during the first year of life. Premature closure of the cranial sutures decrease the intracranial volume and space available for the rapidly developing brain. Cranial vault remodeling (CVR) is the current standard of care to mitigate any possible developmental delay secondary to craniosynostosis and also improve the head shape. CVR is a combined surgery between the neurosurgeon who takes off the cranial bone/bones, and the craniofacial surgeon who assists and reconstructs the cranium with absorbable plates and screws.

After surgery, although there is no doubt that there is an improvement in head shape, the craniofacial skeleton and the soft tissues, but there is less data, and virtually no functional imaging information available addressing the effect of CVR surgery on the growing brain.

The main objective of this project would be to begin to explore the relationship of CVR and it requisite effects on the growing brain with a cohort of patients who are set to undergo CVR, while performing a battery of neurodevelopmental and imaging studies pre- and post-operatively and compare with normative controls. This is one part of a three-center study collaborating with craniofacial units at Yale University and Wake Forest University in which similar, if not identical protocols will be carried out. We hope that analyses of these data will provide better insight into and greater definition of the effect of CVR and the secondarily available increase in intra-cranial volume on the growing brain in the clinical setting of craniosynostosis.

ELIGIBILITY:
Inclusion Criteria:

* Up to 500 children, for all subjects, age of initial study entry: one test group between 3-6 months old( endoscopic assisted) , and the other 6-24 months of age ( open CVR) ) once enrolled, children will be included until 4 years of age.
* Diagnosed with craniosynostosis, single or multiple suture
* Babies with craniosynostosis syndrome including but not limited to Pfieffers, Aperts, Crouzons,and Menkes.
* Approximately 60 age-matched controls (3 in each group) not diagnosed with craniosynostosis syndrome, stratified by age groups starting at 3 months, 5 months, 7 months, 9 month 11 months, 13 months, 15 months, 17 months, 19 months, then every 3 months, 22 months, 25 months, 28 months, 31 months, 34 months, 37 months,40 months,43 months,46 months,49 months.

Exclusion Criteria:

* Children not meeting the inclusion criteria
* Children with traumatic brain injury, brain cancer, or VP shunt that could affect development.
* Children who have already undergone CVR repair
* Developmentally Normal children who cannot undergo or cannot be still for an awake or asleep non-sedated MRI

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of brain development via diagnostic imaging | From 2 months age to 4 years of age
  Will establish pilot data to establish a normative curve of white-matter tract development in normal children under 4 years of age using (DTI). Fractional anisotropy (FA) (a main DTI parameter sensitive to white matter integrity) maps will be created to achieve a normative "white matter change curve" with from infancy to pre-school age.
Assessment of the change in white matter tract organization after cranial vaut remodeling surgery (CVR) | From 2 months age to 4 years of age
  Will quantify the change in white matter tract organization after cranial vault remodeling (CVR) surgery in patients with craniosynostosis by analyzing pre- and post-operative DTI data. This experimental cohort will also be examined in comparison to age-matched controls, pooled with other centers and compared with published data sets of normal babies from the Baby Connectome Project. . The imaging will be repeated at three intervals after surgery leading up to approximately 4 years of age.

SECONDARY OUTCOMES:
Assessment of neurodevelopmental test results in craniosynostosis patients | From 2 months of age to 4 years of age
  Will assess neurodevelopmental test results in craniosynostosis patients and seek to correlate these findings with white matter tract changes

CONTACTS AND LOCATIONS:
Overall Officials: Eylem Ocal, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States